CLINICAL TRIAL: NCT00753051
Title: Treatment of Clozapine-resistant Schizophrenia : Comparison Between Augmentation With Haloperidol and Electroconvulsive Therapy
Brief Title: Treat Clozapine ( CLZ )-Resistant Schizophrenia Comparing CLZ + Haloperidol vs. CLZ + Electroconvulsive Therapy (ECT)
Acronym: TCRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Suchat Paholpak, Professor Doctor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE501122
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Schizophrenia
Keywords: clozapine-resistant schizophrenics; haloperidol augmenting clozapine; electroconvulsive therapy augmenting clozapine
MeSH Terms: conditions — Schizophrenia | interventions — Haloperidol; Clozapine; Electroconvulsive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. (Active Comparator): clozapine as the main agent and it will be adjuncted by haloperidol
  Interventions: Drug: clozapine+haloperidol
- 2. (Active Comparator): clozapine as the main agent and it will be adjuncted by electroconvulsive therapy
  Interventions: Drug: clozapine,electroconvulsive therapy

INTERVENTIONS:
Drug: clozapine+haloperidol — clozapine 300-900 mg/d haloperidol 4-60 mg/d
  Other Names: clopaze, haloperidol
  Arms: 1.
Drug: clozapine,electroconvulsive therapy — clozapine 300-900 mg/d electroconvulsive therapy 4-12 times
  Other Names: clopaze , Thymatron ECT machine
  Arms: 2.

SUMMARY:
Clozapine treatment resistant schizophrenia is still prevalent.The effectiveness of augmenting clozapine : one augmenting with haloperidol and the other with electroconvulsive therapy should be determined.This study is a randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

1. schizophrenic patients diagnosed with schedules for clinical assessment in neuropsychiatry ( SCAN )in accordance with DSM-IV-TR or ICD-10
2. Resistant to at least 6 weeks of clozapine treatment in therapeutic dosage
3. Voluntary to participate the research protocol expressed by signing informed consent form

Exclusion Criteria:

1. Patient does not volunteer himself or herself
2. Patient is having epilepsy, DM, cardiac disease, autistic disorder and illiterate
3. Patient is deaf, blind , dumb to obstruct good communication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-06; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
PANSS , HAM-D , CGI , AIMS Scores | every 4 weeks for 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Suchat Paholpak, MD, Principal Investigator — Department of Psychiatry.Faculty of Medicine.Khon Kaen University
Locations (1):
- Department of Psychiatry.Faculty of Medicine.KhonKaen University., Muang, KhonKaen, Thailand